CLINICAL TRIAL: NCT01336465
Title: Phase II Randomized Double-Blind Placebo-Controlled Study to Evaluate the Efficacy and Safety of rhuMAb Beta7 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Evaluate the Efficacy and Safety of rhuMAb Beta7 in Patients With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABS4986g; GP27778 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- rhuMAb Beta7 (Experimental)
  Interventions: Drug: rhuMAb Beta7
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Repeating subcutaneous injection
  Arms: placebo
Drug: rhuMAb Beta7 — Repeating subcutaneous injection
  Arms: rhuMAb Beta7

SUMMARY:
This Phase II study is a randomized, double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of rhuMAb Beta7 in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe ulcerative colitis outpatient
* Disease duration at time of screening of >/= 12 weeks

Exclusion Criteria:

* Extensive colonic resection or subtotal or total colectomy
* Presence of an ileostomy or colostomy
* Moderate to severe anemia
* A history or evidence of colonic mucosal dysplasia
* Pregnant or lactating
* Significant uncontrolled co-morbidity, such as neurological, cardiac, pulmonary, renal, hepatic, endocrine, or gastrointestinal (GI) disorders
* Significant screening ECG abnormalities, including evidence of acute myocardial infarction, complete left bundle branch block, second-degree heart block, or complete heart block
* Poorly controlled diabetes
* Impaired renal function
* Impaired hepatic function in the absence of a diagnosis of primary sclerosing cholangitis
* Positive tests for antibodies indicating active or prior infection with HIV or hepatitis B (HBV) or C (HCV)
* Positive screening test for latent mycobacterium tuberculosis (TB) infection
* Demyelinating disease
* Received any investigational treatment within 12 weeks prior to initiation of study treatment
* Previous exposure to rhuMAb Beta7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical remission defined as a Mayo Clinic Score (MCS) </= 2 with no individual subscore exceeding 1 point | Week 10

SECONDARY OUTCOMES:
Clinical response as defined by at least a 3-point decrease and 30% reduction from baseline in MCS and a >/=1-point decrease in rectal bleeding subscore or absolute rectal bleeding score of 0 or 1 | Week 6 and Week 10
Clinical remission defined by a MCS </= 2 with no individual subscore exceeding 1 point | Week 6
Proportion of patients with endoscopic score and rectal bleeding score of 0 | Week 6 and Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Sharon O'Byrne, M.D., Study Director — Genentech, Inc.
Locations (46):
- United States (8):
  - San Diego, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Chevy Chase, Maryland
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - Great Neck, New York
  - Cincinnati, Ohio
- Australia (5):
  - Garran, Australian Capital Territory
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
- Belgium (4):
  - Bonheiden
  - Ghent
  - Leuven
  - Liège
- Canada (3):
  - Edmonton, Alberta
  - London, Ontario
  - Woodbridge, Ontario
- Czechia (4):
  - Hradec Králové
  - Náchod
  - Ostrava - Poruba
  - Zlín
- Germany (5):
  - Berlin
  - Hanover
  - Kiel
  - Minden
  - Ulm
- Hungary (4):
  - Budapest
  - Gyöngyös
  - Győr
  - Mosonmagyaróvár
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- New Zealand (4):
  - Auckland
  - Christchurch
  - Dunedin
  - Takapuna
- Barcelona, Barcelona, Spain
- United Kingdom (3):
  - Harrow
  - London
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Vermeire S, O'Byrne S, Keir M, Williams M, Lu TT, Mansfield JC, Lamb CA, Feagan BG, Panes J, Salas A, Baumgart DC, Schreiber S, Dotan I, Sandborn WJ, Tew GW, Luca D, Tang MT, Diehl L, Eastham-Anderson J, De Hertogh G, Perrier C, Egen JG, Kirby JA, van Assche G, Rutgeerts P. Etrolizumab as induction therapy for ulcerative colitis: a randomised, controlled, phase 2 trial. Lancet. 2014 Jul 26;384(9940):309-18. doi: 10.1016/S0140-6736(14)60661-9. Epub 2014 May 9. PMID 24814090